CLINICAL TRIAL: NCT04527692
Title: Exploring the Quality of Life of Children/Adolescents in Palliative Settings and That of Their Parents
Brief Title: Quality of Life of Children/Adolescents in Palliative Care Settings
Acronym: MOSAIK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/19/0347; 2019-A02315-52 (Other: ID-RCB)
Record Dates: First submitted 2020-07-29; First posted 2020-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Palliative Care
Keywords: child; parents; quality of life
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Child: Children/adolescents from 1 to 18 years of age with a serious illness requiring follow-up by a regional pediatric palliative care resource team and/or temporarily hospitalized.
  Interventions: Other: Questionnaire
- Parents: Adult person with parental authority over a child between the ages of 1 and 18 who is a carrier of a serious illness and requires follow-up by a regional pediatric palliative care resource team and/or is temporarily hospitalized.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — semi-structured interviews on the quality of life

SUMMARY:
Investigators will propose to each family monitored by the teams to participate in the study (children between 1 and 18 years old, families understanding and speaking a minimum of French).

Semi-directed interviews are organized with children/adolescents and their parents who have agreed to participate in the study. The interviews are conducted by the care teams themselves. Socio-demographic data are collected.

DETAILED DESCRIPTION:
An information letter will be distributed to the children and parents and their non opposition to their participation will be sought (or assent for the child via a written document adapted to the age) will be systematically requested.

Several instruments will be used by the members of the paediatric teams during their routine home or hospital visits to children and their families: the CPOS (Downing 2018), the KINDL (generic questionnaire on quality of life validated for healthy children, Erhart et al. 2009), the QOLLTI-F v.2 (questionnaire on quality of life for parents, Cohen 2007, 2015).

The interviews will therefore be semi-directed interviews with children/adolescents and their parents who have agreed to participate in the study. The interviews will be conducted by the care teams themselves. In addition to the CPOS, KINDL and QOOLTI-F, socio-demographic data are collected.

ELIGIBILITY:
Inclusion Criteria:

* Children/adolescents aged 1 to 18 years with a serious illness and requiring follow-up by a regional pediatric palliative care resource team and/or temporarily hospitalized.
* Having given his non-opposition to his participation.
* A minor of whom at least one of the two holders of parental authority has given his or her consent to the participation of their child.
* Child of whom one of the two holders of parental authority has himself agreed to participate in the study.

Exclusion Criteria:

* Children/adolescents at the end of life (imminent death foreseeable).
* Children/adolescents and their parents who do not understand French.
* Child or parent under legal protection (guardianship, curatorship).

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Child/parent pair agrees to participate, they give their agreement orally and their non-opposition is documented in the patient's medical record.
  Interviews are conducted at home and/or at the hospital depending on where the child is usually cared for by the usual care team.
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-12-15 (Estimated); Study Completion 2022-11-15 (Estimated)

PRIMARY OUTCOMES:
Quality of life measure | Day 1
  Exploring the quality of life of children/adolescents in palliative settings and that of their parents through the development of the Childrens palliative outcome scale.

SECONDARY OUTCOMES:
psychometric measure - KINDL | Day 1
  using the validated questionnaire KINDL, French version
psychometric measure - QOLLTI-F | Day 1
  using the the validated questionnaire Quality of life in life threatening illness-family caregiver QOLLTI-F.
psychometric measure - Children's palliative outcome scale | Day 1
  Documentation of the psychometric properties of the Children's palliative outcome scale

CONTACTS AND LOCATIONS:
Overall Officials: Agnes SUC, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Agnès SUC, Toulouse, France

IPD SHARING:
Plan to Share IPD: No